CLINICAL TRIAL: NCT05666336
Title: Proteomics Combined With Metabolomics Studies on the Efficacy of Telitacicept in Chinese Patients of Systemic Lupus Erythematosus
Brief Title: Multi-omics Studies on the Efficacy of Telitacicept in Chinese SLE Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fen Li (Other)
Responsible Party: Sponsor-Investigator, Fen Li, chief physician, Central South University
Organization: Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYF2022151
Record Dates: First submitted 2022-12-08; First posted 2022-12-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Telitacicept; efficiency; omics
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept; Hydroxychloroquine; Prednisone; prednylidene; Methylprednisolone; Cyclophosphamide; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): The treatment regimen consists of four drugs, a glucocorticoid plus Telitacicept plus hydroxychloroquine plus an immunosuppressor.
  Prednisone(30mg, Qd) or Methylprednisolone(24mg, Qd) plus Telitacicept(160mg, Qw) plus Hydroxychloroquine (0.2g, Qd) plus cyclophosphamide(0.8g, Qm) or Mycophenolate Mofetil (0.5g, Bid) or Tacrolimus (1mg, Bid) The above treatment will continue for 24 weeks.
  Interventions: Biological: Telitacicept; Drug: Hydroxychloroquine; Drug: Prednisone; Drug: Methylprednisolone; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Biological: Telitacicept — It is necessary and will be given by subcutaneous injection of 160mg/week for 24 weeks.
  Other Names: RC18
Drug: Hydroxychloroquine — It is necessary and will be given by oral administration of 0.2g/day for 24 weeks.
  Other Names: HCQ
Drug: Prednisone — It is permitted which can be interchangeable with methylprednisolone. It will be given by oral administration of 30mg/day from beginning and be lowed dosage during the treatment of 24 weeks.
  Other Names: PRED
Drug: Methylprednisolone — It is permitted which can be interchangeable with prednisone. It will be given by oral administration of 24mg/day from beginning and be lowed dosage during the treatment of 24 weeks.
  Other Names: MP
Drug: Cyclophosphamide — It is permitted which can be interchangeable with mycophenolate mofetil or tacrolimus. It will be given by oral administration of 0.8g/month for 24 weeks.
  Other Names: CTX
Drug: Mycophenolate Mofetil — It is permitted which can be interchangeable with cyclophosphamide or tacrolimus. It will be given by oral administration of 0.5g twice a day for 24 weeks.
  Other Names: MMF
Drug: Tacrolimus — It is permitted which can be interchangeable with cyclophosphamide or mycophenolate mofetil. It will be given by oral administration of 1mg twice a day for 24 weeks.
  Other Names: TAC

SUMMARY:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disease with abnormal activation of B lymphocytes, which may result in many adverse consequences and even death if not treated actively. Telitacicept, approved conditionally in China in March 2021, is a biologic agent targeting B lymphocyte stimulator (BLyS）and a proliferating inducing ligand (APRIL) dually for patients with active SLE patients who have not responded to conventional treatment. The investigators hope to screen predictive biomarkers of efficacy and explore the mechanism of difference in efficacy of Telitacicept with Chinese characteristics by omics.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disease with abnormal activation of B lymphocytes, which may result in many adverse consequences and even death if not treated actively. Due to the poor therapeutic efficacy and prominent adverse reactions after long-term use of glucocorticoid combined immunosuppressants, the development of targeted drug use for SLE has become a hot area of research for several years. Telitacicept, approved conditionally in China in March 2021, is a biologic agent targeting B lymphocyte stimulator (BLyS）and a proliferating inducing ligand (APRIL) dually for patients with active SLE patients who have not responded to conventional treatment. As another important part of targeted drug use, the research on biomarkers predictive of drug response is also in full swing in the treatment of SLE. The omics technology has unique advantages in screening biomarkers and exploring the mechanism of drug action. The integrated analysis of multi omics can mutually verify and supplement the screening results of a single omics, so as to more systematically and comprehensively analyze the biological molecular functions and regulatory mechanisms. Therefore, this topic selects serum proteomics combined with metabolomics to screen biomarkers for the prediction of the efficacy of Telitacicept, and to explore the mechanism of the difference in the efficacy of Telitacicept, with a view to providing meaningful reference for the exploration of SLE precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of SLE according to American College of Rheumatology (ACR) classification criteria 1997 and clinically active disease.
2. Patients with good compliance, will sign the informed consent before the test.
3. Patients who have received conventional treatment for SLE, and the type and dose of treatment drugs have been stable for at least 30 days.
4. Patients who have a positive anti-nuclear antibody test result and SELENA-SLEDAI score ≥8 at screening. If there is a low complement and/or positive anti-dsDNA antibody, the SELENA-SLEDAI score can be defined as ≥ 6 points.

Exclusion Criteria:

1. Patients with severe lupus nephritis, defined as urinary protein > 6g /24 hours or serum creatinine > 221μmol/L within the last 2 months, or who require hemodialysis.
2. Patients with SLE-caused or non-SLE-caused central nervous system disease within the last 2 months.
3. Patients with severe condition in blood, important organs including heart, liver, gastrointestinal tract and endocrine system which are not related with SLE.
4. Patients who use prednisone ≥100mg/d over 14 days or receive plasma replacement and suffer from active infection within the last 1 month.
5. Patients who received any other targeted agents over the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
SLE Responder Index (SRI) 4 response rate | week 24
  (1) Definition of SRI4: ≥4 point reduction from baseline in SELENA-SLEDAI score, no worsening (<0.3 point increase from baseline) in Physician's Global Assessment (PGA) and no new British Isles Lupus Assessment Group (BILAG) A organ domain score or two new BILAG B organ domain scores vs baseline. (2) The patients acquired SRI4 were classified as Good Responders (GR), The patients not acquired SRI4 were classified as Non-Responders (NR).

SECONDARY OUTCOMES:
The changes of glucocorticoids dose | week 24
  The percentage of patients whose average prednisone dose was ≤7.5 mg/day or reduced by ≥25% from baseline.
The variation of serum markers | week 24
  The variation of serum markers including BLyS,APRIL,CD19+B lymphocytes count, anti-dsDNA antibodies, IgG, IgA, IgM, complement3(C3), and complement4(C4) at baseline and after 24 weeks' treatment.
Proteomics | week 24
  Screening and comparison of different proteins
Metabonomics | week 24
  Screening and comparison of different metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Fen Li, doctor, Principal Investigator — Central South University
Locations (1):
- Department of Rheumatology and Immunology, Xiangya Second Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhillon S. Telitacicept: First Approval. Drugs. 2021 Sep;81(14):1671-1675. doi: 10.1007/s40265-021-01591-1. PMID 34463932
- [Background] Fan Y, Gao D, Zhang Z. Telitacicept, a novel humanized, recombinant TACI-Fc fusion protein, for the treatment of systemic lupus erythematosus. Drugs Today (Barc). 2022 Jan;58(1):23-32. doi: 10.1358/dot.2022.58.1.3352743. PMID 35107091
- [Background] Hruskova Z, Tesar V. Lessons learned from the failure of several recent trials with biologic treatment in systemic lupus erythematosus. Expert Opin Biol Ther. 2018 Sep;18(9):989-996. doi: 10.1080/14712598.2018.1504918. Epub 2018 Jul 31. PMID 30040494
- [Background] Merrill JT, Neuwelt CM, Wallace DJ, Shanahan JC, Latinis KM, Oates JC, Utset TO, Gordon C, Isenberg DA, Hsieh HJ, Zhang D, Brunetta PG. Efficacy and safety of rituximab in moderately-to-severely active systemic lupus erythematosus: the randomized, double-blind, phase II/III systemic lupus erythematosus evaluation of rituximab trial. Arthritis Rheum. 2010 Jan;62(1):222-33. doi: 10.1002/art.27233. PMID 20039413
- [Background] Vital EM, Dass S, Buch MH, Henshaw K, Pease CT, Martin MF, Ponchel F, Rawstron AC, Emery P. B cell biomarkers of rituximab responses in systemic lupus erythematosus. Arthritis Rheum. 2011 Oct;63(10):3038-47. doi: 10.1002/art.30466. PMID 21618204
- [Background] Pirone C, Mendoza-Pinto C, van der Windt DA, Parker B, O Sullivan M, Bruce IN. Predictive and prognostic factors influencing outcomes of rituximab therapy in systemic lupus erythematosus (SLE): A systematic review. Semin Arthritis Rheum. 2017 Dec;47(3):384-396. doi: 10.1016/j.semarthrit.2017.04.010. Epub 2017 May 5. PMID 28602359
- [Background] Cecchi I, Perez-Sanchez C, Sciascia S, Radin M, Arias de la Rosa I, Barbarroja Puerto N, Scudeler L, Perez-Sanchez L, Patino Trives AM, Aguirre Zamorano MA, Menegatti E, Roccatello D, Lopez-Pedrera C. Circulating microRNAs as potential biomarkers for monitoring the response to in vivo treatment with Rituximab in systemic lupus erythematosus patients. Autoimmun Rev. 2020 Apr;19(4):102488. doi: 10.1016/j.autrev.2020.102488. Epub 2020 Feb 13. No abstract available. PMID 32062026
- [Background] Davies JC, Midgley A, Carlsson E, Donohue S, Bruce IN, Beresford MW, Hedrich CM. Urine and serum S100A8/A9 and S100A12 associate with active lupus nephritis and may predict response to rituximab treatment. RMD Open. 2020 Jul;6(2):e001257. doi: 10.1136/rmdopen-2020-001257. PMID 32723832
- [Background] Davies JC, Carlsson E, Midgley A, Smith EMD, Bruce IN, Beresford MW, Hedrich CM; BILAG-BR and MRC MASTERPLANS Consortia. A panel of urinary proteins predicts active lupus nephritis and response to rituximab treatment. Rheumatology (Oxford). 2021 Aug 2;60(8):3747-3759. doi: 10.1093/rheumatology/keaa851. PMID 33313921
- [Background] Iaccarino L, Andreoli L, Bocci EB, Bortoluzzi A, Ceccarelli F, Conti F, De Angelis R, De Marchi G, De Vita S, Di Matteo A, Emmi G, Emmi L, Gatto M, Gerli R, Gerosa M, Govoni M, Larosa M, Meroni PL, Mosca M, Pazzola G, Reggia R, Saccon F, Salvarani C, Tani C, Zen M, Frigo AC, Tincani A, Doria A. Clinical predictors of response and discontinuation of belimumab in patients with systemic lupus erythematosus in real life setting. Results of a large, multicentric, nationwide study. J Autoimmun. 2018 Jan;86:1-8. doi: 10.1016/j.jaut.2017.09.004. Epub 2017 Sep 19. PMID 28935492
- [Background] Piantoni S, Regola F, Masneri S, Merletti M, Lowin T, Airo P, Tincani A, Franceschini F, Andreoli L, Pongratz G. Characterization of B- and T-Cell Compartment and B-Cell Related Factors Belonging to the TNF/TNFR Superfamily in Patients With Clinically Active Systemic Lupus Erythematosus: Baseline BAFF Serum Levels Are the Strongest Predictor of Response to Belimumab after Twelve Months of Therapy. Front Pharmacol. 2021 May 21;12:666971. doi: 10.3389/fphar.2021.666971. eCollection 2021. PMID 34093196
- [Background] Yao X, Ren Y, Zhao Q, Chen X, Jiang J, Liu D, Hu P. Pharmacokinetics analysis based on target-mediated drug distribution for RC18, a novel BLyS/APRIL fusion protein to treat systemic lupus erythematosus and rheumatoid arthritis. Eur J Pharm Sci. 2021 Apr 1;159:105704. doi: 10.1016/j.ejps.2021.105704. Epub 2021 Jan 10. PMID 33440243
- [Background] Gordon C, Wofsy D, Wax S, Li Y, Pena Rossi C, Isenberg D. Post Hoc Analysis of the Phase II/III APRIL-SLE Study: Association Between Response to Atacicept and Serum Biomarkers Including BLyS and APRIL. Arthritis Rheumatol. 2017 Jan;69(1):122-130. doi: 10.1002/art.39809. Epub 2016 Dec 2. PMID 27390168
- [Background] Merrill JT, Wallace DJ, Wax S, Kao A, Fraser PA, Chang P, Isenberg D; ADDRESS II Investigators. Efficacy and Safety of Atacicept in Patients With Systemic Lupus Erythematosus: Results of a Twenty-Four-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase IIb Study. Arthritis Rheumatol. 2018 Feb;70(2):266-276. doi: 10.1002/art.40360. PMID 29073347
- [Background] Stohl W, Hilbert DM. The discovery and development of belimumab: the anti-BLyS-lupus connection. Nat Biotechnol. 2012 Jan 9;30(1):69-77. doi: 10.1038/nbt.2076. PMID 22231104
- [Background] Shu W, Guan S, Yang X, Liang L, Li J, Chen Z, Zhang Y, Chen L, Wang X, Huang M. Genetic markers in CYP2C19 and CYP2B6 for prediction of cyclophosphamide's 4-hydroxylation, efficacy and side effects in Chinese patients with systemic lupus erythematosus. Br J Clin Pharmacol. 2016 Feb;81(2):327-40. doi: 10.1111/bcp.12800. Epub 2015 Dec 25. PMID 26456622
- [Background] McBride JM, Jiang J, Abbas AR, Morimoto A, Li J, Maciuca R, Townsend M, Wallace DJ, Kennedy WP, Drappa J. Safety and pharmacodynamics of rontalizumab in patients with systemic lupus erythematosus: results of a phase I, placebo-controlled, double-blind, dose-escalation study. Arthritis Rheum. 2012 Nov;64(11):3666-76. doi: 10.1002/art.34632. PMID 22833362
- [Background] Kalunian KC, Merrill JT, Maciuca R, McBride JM, Townsend MJ, Wei X, Davis JC Jr, Kennedy WP. A Phase II study of the efficacy and safety of rontalizumab (rhuMAb interferon-alpha) in patients with systemic lupus erythematosus (ROSE). Ann Rheum Dis. 2016 Jan;75(1):196-202. doi: 10.1136/annrheumdis-2014-206090. Epub 2015 Jun 2. PMID 26038091
- [Background] Vasquez-Canizares N, Wahezi D, Putterman C. Diagnostic and prognostic tests in systemic lupus erythematosus. Best Pract Res Clin Rheumatol. 2017 Jun;31(3):351-363. doi: 10.1016/j.berh.2017.10.002. Epub 2017 Nov 6. PMID 29224677
- [Background] Pedrosa L, Fernandez-Miranda I, Perez-Callejo D, Quero C, Rodriguez M, Martin-Acosta P, Gomez S, Gonzalez-Rincon J, Santos A, Tarin C, Garcia JF, Garcia-Arroyo FR, Rueda A, Camacho FI, Garcia-Cosio M, Heredero A, Llanos M, Mollejo M, Piris-Villaespesa M, Gomez-Codina J, Yanguas-Casas N, Sanchez A, Piris MA, Provencio M, Sanchez-Beato M. Proposal and validation of a method to classify genetic subtypes of diffuse large B cell lymphoma. Sci Rep. 2021 Jan 21;11(1):1886. doi: 10.1038/s41598-020-80376-0. PMID 33479306
- [Background] Zhang X, Jin M, Wu H, Nadasdy T, Nadasdy G, Harris N, Green-Church K, Nagaraja H, Birmingham DJ, Yu CY, Hebert LA, Rovin BH. Biomarkers of lupus nephritis determined by serial urine proteomics. Kidney Int. 2008 Sep;74(6):799-807. doi: 10.1038/ki.2008.316. Epub 2008 Jul 2. PMID 18596723
- [Background] Parra S, Heras M, Herrero P, Amigo N, Garces E, Girona J, Correig X, Canela N, Castro A. Gelsolin: a new biomarker of disease activity in SLE patients associated with HDL-c. Rheumatology (Oxford). 2020 Mar 1;59(3):650-661. doi: 10.1093/rheumatology/kez293. PMID 31504936
- [Background] Troyer B, Rodgers J, Wolf BJ, Oates JC, Drake RR, Nowling TK. Glycosphingolipid Levels in Urine Extracellular Vesicles Enhance Prediction of Therapeutic Response in Lupus Nephritis. Metabolites. 2022 Feb 1;12(2):134. doi: 10.3390/metabo12020134. PMID 35208209
- [Background] Romick-Rosendale LE, Brunner HI, Bennett MR, Mina R, Nelson S, Petri M, Kiani A, Devarajan P, Kennedy MA. Identification of urinary metabolites that distinguish membranous lupus nephritis from proliferative lupus nephritis and focal segmental glomerulosclerosis. Arthritis Res Ther. 2011;13(6):R199. doi: 10.1186/ar3530. Epub 2011 Dec 7. PMID 22152586
- [Background] Guleria A, Phatak S, Dubey D, Kumar S, Zanwar A, Chaurasia S, Kumar U, Gupta R, Aggarwal A, Kumar D, Misra R. NMR-Based Serum Metabolomics Reveals Reprogramming of Lipid Dysregulation Following Cyclophosphamide-Based Induction Therapy in Lupus Nephritis. J Proteome Res. 2018 Jul 6;17(7):2440-2448. doi: 10.1021/acs.jproteome.8b00192. Epub 2018 Jun 18. PMID 29877087
- [Background] Tanaka Y, Kubo S, Miyagawa I, Iwata S, Nakayamada S. Lymphocyte phenotype and its application to precision medicine in systemic autoimmune diseases✰. Semin Arthritis Rheum. 2019 Jun;48(6):1146-1150. doi: 10.1016/j.semarthrit.2019.04.007. Epub 2019 Apr 25. PMID 31079846